CLINICAL TRIAL: NCT04354844
Title: Quality of Life in Cardiac Patients Attending Assuit University Children Hospital
Brief Title: Quality of Life in Cardiac Pediatric Patients Attending Assuit Univeristy Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nardeen Emad Elway, principal investigator, Assiut University
Other Study IDs: qolicp
Record Dates: First submitted 2020-04-09; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Quality of Life
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cyanotic and acyanotic group: questinnaire
  Interventions: Behavioral: questionnaire

INTERVENTIONS:
Behavioral: questionnaire — questionnaire

SUMMARY:
Quality of life(QOL) is defined as the individual perception related with their state in life in terms of the cultural structure and system of values in which they live. Their objectives, expectations, standards and concerns, whereas health related quality of life is defined as the patient subjective perception of the impact of their disease or its treatment.(1) Cardiac disease is the most common congenital defect in children, with an incidence of eight in every 1000 live births. Multiple factors have improved and prolonged the lives of children and adolescents with congenital heart disease over the last few decades(2)

DETAILED DESCRIPTION:
Quality of life(QOL) is defined as the individual perception related with their state in life in terms of the cultural structure and system of values in which they live. Their objectives, expectations, standards and concerns, whereas health related quality of life is defined as the patient subjective perception of the impact of their disease or its treatment.(1) Cardiac disease is the most common congenital defect in children, with an incidence of eight in every 1000 live births. Multiple factors have improved and prolonged the lives of children and adolescents with congenital heart disease over the last few decades(2) Diagnosis of a life-threatening illness during a child's formative years can have far-reaching effects that ripple through the family and across a lifetime. Infants with complex CHD experience a range of uncommon and painful events, such as separation from their mother at birth, urgent transfer to specialized intensive care, frequent invasive medical procedures, feeding difficultiesand withdrawal from narcotic pain relief. These earlylife experiences can have profound consequences for the developing child, shaping brain development, the body's immune system and responses to stress.(5) From a neurodevelopmental perspective, children with CHD experience greater difficulties compared with their healthy peers. The risk and severity of neurodevelopmental impairment increases with greater CHD complexity, the presence of a genetic disorder or syndrome, and greater psychological stress. During infancy, the most pronounced difficulties occur in motor functioning. By early childhood, studies show that children with complex CHD have an increased risk of neurodevelopmental impairment, in fine and gross motor skills, and language, attention, executive functioning, emotion regulation and behaviour.(7)

ELIGIBILITY:
Inclusion Criteria:

* - Infants of both sex.
* Age :from 2 years to 18 years.
* Attending Assuit University Children Hospital including NICU, pediatric cardiology department, outpatient clinics.
* Patients diagnosed with congenital heart disease (cyanotic, acyanotic, cardiomyopathy, rheumatic heart).

Exclusion Criteria:

* - patients suspected to have congenital heart but excluded on echo diagnosis. patient with any associated lesions (patients have any congenital anomalies with congenital heart like down syndrome)

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Infants of both sex.
  * Age :from day one to 18 years.
  * Attending Assuit University Children Hospital including NICU, pediatric cardiology department, outpatient clinics.
  * Patients diagnosed with congenital heart disease (cyanotic, acyanotic, cardiomyopathy, rheumatic heart).
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate quality of life in cardiac pediatric patients | 1 year
  Questionnaire

SECONDARY OUTCOMES:
How to improve quality of life in all cardiac pediatric patients and their families | 1year
  Questionnaire

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Davis CC, Brown RT, Bakeman R, Campbell R. Psychological adaptation and adjustment of mothers of children with congenital heart disease: stress, coping, and family functioning. J Pediatr Psychol. 1998 Aug;23(4):219-28. doi: 10.1093/jpepsy/23.4.219. PMID 9718895
- [Background] Gee DG, Gabard-Durnam LJ, Flannery J, Goff B, Humphreys KL, Telzer EH, Hare TA, Bookheimer SY, Tottenham N. Early developmental emergence of human amygdala-prefrontal connectivity after maternal deprivation. Proc Natl Acad Sci U S A. 2013 Sep 24;110(39):15638-43. doi: 10.1073/pnas.1307893110. Epub 2013 Sep 9. PMID 24019460
- [Background] Marino BS, Lipkin PH, Newburger JW, Peacock G, Gerdes M, Gaynor JW, Mussatto KA, Uzark K, Goldberg CS, Johnson WH Jr, Li J, Smith SE, Bellinger DC, Mahle WT; American Heart Association Congenital Heart Defects Committee, Council on Cardiovascular Disease in the Young, Council on Cardiovascular Nursing, and Stroke Council. Neurodevelopmental outcomes in children with congenital heart disease: evaluation and management: a scientific statement from the American Heart Association. Circulation. 2012 Aug 28;126(9):1143-72. doi: 10.1161/CIR.0b013e318265ee8a. Epub 2012 Jul 30. PMID 22851541